CLINICAL TRIAL: NCT03026946
Title: Efficacy of Oral Alitretinoin Versus Oral Cyclosporine in Patients With Severe Recurrent Vesicular Hand Eczema. A Randomized Prospective Open-label Trial With Blinded Outcome Assessment
Brief Title: Alitretinoin vs Cyclosporine in Severe Recurrent Vesicular Hand Eczema
Acronym: ALICsA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Marie-Louise A Schuttelaar, MD, PhD, MD, PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 54659
Record Dates: First submitted 2016-12-13; First posted 2017-01-20 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Hand Eczema
Keywords: Alitretinoin; Cyclosporine A; Hand eczema
MeSH Terms: interventions — Alitretinoin; Cyclosporine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alitretinoin (Active Comparator): Patients with severe recurrent vesicular hand eczema, randomized to treatment with alitretinoin.
  Interventions: Drug: Alitretinoin
- Cyclosporin A (Active Comparator): Patients with severe recurrent vesicular hand eczema, randomized to treatment with cyclosporin A.
  Interventions: Drug: cyclosporin A

INTERVENTIONS:
Drug: Alitretinoin — Oral alitretinoin capsule of 30mg once daily for a total of 24 weeks.
  Other Names: Toctino; 9-cis-retinoic acid; ATC code: D11AH04
  Arms: Alitretinoin
Drug: cyclosporin A — Oral cyclosporine A start dose 5 mg/kg/day (split in 2 doses), decreasing the dose after 8 weeks to 3 - 3.5 mg/kg/day (split in 2 doses). The treatment period is 24 weeks.
  Other Names: Neoral
  Arms: Cyclosporin A

SUMMARY:
The purpose of this study is to compare the efficacy of alitretinoin and cyclosporine in the treatment of patients with severe recurrent vesicular hand eczema.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years and ≤ 75 years

* Severe or very severe recurrent vesicular hand eczema for a minimum duration of 3 months as defined by a Physician Global Assessment (PGA) using a validated Photoguide
* Refractory to standard therapy, defined as:

Patients received treatment with topical corticosteroids of class II or higher for at least 8 weeks within 3 months before enrolment, with either no response or a transient response. Patients had also received standard skin care, including emollients and barrier protection as appropriate, without significant improvement. Patients had avoided irritants and contact allergens, if identified, without significant improvement.

* Women of childbearing potential are required to use at least two forms of contraception for at least 1 month before starting treatment, during treatment, and for at least 1 month after finishing treatment; these women are required to take monthly pregnancy tests
* Able to provide written Informed Consent
* Able to speak and read the Dutch language

Exclusion Criteria:

General criteria prior to randomization

* Treated with alitretinoin or cyclosporine in the previous 3 months
* Other morphologic types of hand eczema as defined by the Danish Contact Dermatitis Group
* Patients with predominantly atopic dermatitis, in which the hands are also involved. (Patients with controlled atopic dermatitis, in which the hands are mainly affected, are eligible for inclusion.)
* Psoriasis of the hands
* Active bacterial, fungal, or viral infection of the hands
* Pregnant/lactating or planning to become pregnant during the study period
* Treatment with systemic medication or UV radiation within the previous 4 weeks
* Mentally incompetent
* Immunocompromised status
* Uncontrolled arterial hypertension (minimally 3 measurements). Systolic pressure > 160 mmHg or diastolic pressure > 95 mmHg, despite starting anti-hypertensive medication (first choice amlodipine 5 mg/day)
* Known or suspected allergy to ingredients in the study medications
* Inclusion in a study of an investigational drug within 60 days prior to start of treatment
* Current malignancy (other than successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and⁄or localized carcinoma in situ of the cervix)
* Current active pancreatitis
* Evidence of alcohol abuse or drug addiction
* Malabsorption
* Currently active gout
* Recurring convulsions / epilepsy
* Living vaccine (including bacillus Calmette-Guérin (BCG), varicella, measles, mumps, rubella, yellow fever, oral polio and oral typhoid) in the last 2 weeks or the planned application of such a vaccine during the study period
* Chronic or recurrent infectious diseases
* Contact sensitizations with clinical relevance to the hands, in which exposure to allergens is not avoided.
* Hypervitaminosis A due to the use of vitamin A supplements containing >2000 IU
* Use of drugs with potential to change the effective dosis of study drugs within the previous 2 weeks Laboratory exclusion criteria post randomization
* Alanine aminotransferase (ALAT) and ⁄or aspartate aminotransferase (ASAT) values > 200% of the upper limit of normal
* Impaired renal function as indicated by a clinically relevant abnormal creatinine value (to be determined by investigator or treating physician)
* Anemia as indicated by a clinically relevant lowered hemoglobin value (to be determined by investigator or treating physician) Alitretinoin specific
* Triglycerides > 200% of the upper limit of normal,
* Cholesterol or low density lipoprotein (LDL) cholesterol values > 200% of the upper limit of normal
* Uncontrolled hypothyroidism (to be determined by investigator or treating physician)

Cyclosporine specific:

* Impaired renal function as indicated by a clinically relevant abnormal creatinine value (to be determined by investigator or treating physician)
* Uremia
* Hyperkalemia
* Hyperuricemia in patients with a medical history of gout

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2017-05-29 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Response to treatment/hand eczema severity (Photoguide) | 24 weeks (end of treatment)

SECONDARY OUTCOMES:
Response to treatment/hand eczema severity (Photoguide) | 12 weeks
Response to treatment/hand eczema severity (Hand Eczema Severity Index, HECSI) | Week 4, 8, 12, 24
Time to response | Week 4, 8, 12, 24
Patient reported improvement (Patient Global Assessment, PaGA) | Week 12 and 24
Safety and tolerability (adverse events) | Up to 24 weeks
Cost-utility. QALY's: registered direct/indirect costs, combined with EQ-5D outcome | Week 12 and 24
Cost-effectiveness: registered direct/indirect costs combined with the primary and secondary effectiveness outcomes (Photoguide/HECSI) | Week 12 and 24
Quality of Life: questionnaire. | Week 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: MLA Schuttelaar, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data will be published anonymously and will not be possible to trace back to individual participants.

REFERENCES:
- [Derived] Oosterhaven JAF, Schuttelaar MLA. Study protocol: efficacy of oral alitretinoin versus oral cyclosporine A in patients with severe recurrent vesicular hand eczema (ALICsA): a randomised prospective open-label trial with blinded outcome assessment. BMJ Open. 2018 Jul 11;8(7):e020192. doi: 10.1136/bmjopen-2017-020192. PMID 29997136